CLINICAL TRIAL: NCT05285683
Title: The Role of Dopamine in the Central Neural Signature of Chronic Pain
Brief Title: The Role of Brain Dopamine in Chronic Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Paul Geha, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00006948
Record Dates: First submitted 2022-02-21; First posted 2022-03-17 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain
Keywords: dopamine; loss of motivation; chronic back pain
MeSH Terms: conditions — Chronic Pain | interventions — Methylphenidate; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Methylphenidate (Active Comparator): 0.5mg/kg
  Interventions: Drug: Methylphenidate
- Carbidopa/levodopa, (Active Comparator): 25mg/100mg
  Interventions: Drug: carbidopa-levodopa
- Placebo (Placebo Comparator): Oral Pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — 0.5 mg/kg
  Arms: Methylphenidate
Drug: carbidopa-levodopa — 25 mg/100 mg
  Arms: Carbidopa/levodopa,
Drug: Placebo — oral pill
  Arms: Placebo

SUMMARY:
Chronic pain is associated with plasticity in the brain limbic system composed mainly of the amygdala, hippocampus, ventral striatum, and cingulate cortex (ACC) /medial prefrontal cortex (mPFC). These brain areas, especially the ventral striatum, receive dopaminergic input from the ventral-tegmental area (VTA). Although there is a significant literature now showing that limbic brain tracks chronic pain intensity and predicts the risk of transition from sub-acute to chronic pain, the role of dopaminergic input to the limbic brain and the change thereof which occurs in chronic pain, is still not clear.

Given the role of dopamine in motivational control and the loss of motivation associated with chronic pain understanding how dopaminergic transmission is altered in the limbic brain of chronic pain patients is critical to the understanding of the pathophysiology of chronic pain. Therefore, the overall aim of this project is to use brain imaging to study how dopaminergic transmission through the oral administration of pro-dopaminergic medications carbidopa/levodopa (CD/LD) and methylphenidate will modulate the brain signature of chronic pain. Chronic pain subjects will be scanned at baseline (no drug administration) and three times after treatment with the two drugs or placebo. The protocol will follow a randomized double-blind approach.

DETAILED DESCRIPTION:
The proposed study is a single center study investigating the effect of dopamine modulation on the brain signature of chronic pain. The patients will undergo 4 scanning visits (baseline, placebo, LD/CD, and MP) the order of the drug visits will be randomized by the investigational drug pharmacy (IDP). In addition, both patients and experimenters will be blind to the intervention given. The patients would have therefore received all the 3 different treatments by the end of the study.

Chronic pain patients will be asked to come to the PI's Lab for 4 visits. On visit 1, after consenting and doing the drug screen, the subject will be asked questions on their pain experience. Subjects will then fill out demographic and clinical questionnaire to assess pain, mood, anxiety, history of early trauma, and stress. Patients will be asked to rate their pain level using a visual analogue scale (VAS).

During visit 1, Dr. Geha will interview patients to inquire about any prior drug allergies including allergy to medications used in this study (Levodopa/Carbidopa and Methylphenidate). Dr. Geha will also explain to the chronic pain patients the possible side effects of LD/CD and MP and hand them a drug information sheet for both medications. Subjects will then undergo 60 minutes of functional and structural scanning, which will serve as a baseline scan.

Visits 2, 3 and 4 for chronic pain patients: Upon arrival, patients will be asked to play Effort Expenditure for Rewards Task (EEfRT) which is a task that assesses motivation. It has been shown to be sensitive to dopaminergic tone in healthy subjects. Before the scan, either the drug (LD/CD or MP) or the placebo will be administered, and patients will wait in the lab for 3 hours and then the EEfRT and scan will be repeated. Pain assessment will occur before and after drug administration. The order (placebo or drug) of the visits will be randomized. Pain assessment will use the VAS and the questionnaires listed below.

* The McGill Pain Questionnaire - Short Form 2 (SF-MPQ-2) is a short-form version of the standard MPQ mentioned above.
* Neuropathic Pain Questionnaire (NPQ) is a 12-item self-report measure used to assess neuropathic pain in adults and discriminate it from non-neuropathic pain. Subjects rate each of the 12 items on a numeric scale from 0 to 100, where 0 indicates no pain and 100 indicates the most extreme pain.
* PainDETECT Questionnaire (PD-Q) is a screening instrument for neuropathic pain comprised on nine items, including a drawing for visual representation of pain. The nine items pertaining to gradation of pain are rated on a 6-point Likert scale where 0=never and 5=very strongly. Pain course pattern and radiating pain domains include visual representations to assist in describing pain.
* Pain Catastrophizing Scale (PCS) is a 13-item self-report measure of negative attitudes towards pain. Responses for each item are presented on a 4-point Likert scale from 0=not at all and 4=all the time.
* Beck Anxiety Index (BAI) is a 21-item self-report measure of severity of anxiety symptoms in the past week. Items are rated on a 4-point Likert scale where 0=not at all and 3=severely, and higher scores indicate greater anxiety symptoms.
* Beck Depression Index (BDI-II) is a 21-item self-report measure of severity of depressive symptoms in the past week. Response choices per item are statements coded numerically from 0-3, where higher values indicate greater impairment.
* Early Trauma Inventory - Self Report (ETI-SR) assesses childhood trauma across 62- items in four domains of traumatic events: general trauma, physical trauma, emotional trauma, and sexual abuse.
* Snaith-Hamilton Pleasure Scale (SHAPS) is a 14-item self-report measure of anhedonia in which subjects are asked to rate their pleasure/enjoyment for each item in the past week on a 4-point Likert scale from 1=definitely agree to 4=definitely disagree, and higher scores indicate higher levels of state anhedonia in the past week.
* Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire consisting of two scales (positive and negative emotions) with 10-items each. Responses to each item are on a 5-point Likert scale from 1=not at all to 5=extremely.
* Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report measure of anxiety and depression for individuals getting outpatient treatment, and responses are scored from 0-3 with higher scores indicating greater levels of anxiety and/or depression.
* CSI Questionnaire is a 25-item self-report measure to determine whether the symptoms of patients is associated with central sensitization (CS). Item responses are on a 4-point scale and can be answered as follows: 0=Never, 1= Rarely, 2=Sometimes, 3=Often and 4=Always. The total score will be used to estimate the severity of central sensitization symptoms.
* Effort Expenditure for Rewards Task (EEfRT) is also a computer-based, multi-trial task. For every trial in the task, subjects are given the opportunity to choose between two different task difficulty levels (hard or easy) to obtain monetary rewards. For all trials, participants made repeated manual button presses within a short period of time. With each press of the button, a virtual 'bar' on the screen raises. Subjects are eligible to win the money for each trial if they can raise the bar to the top of the screen within the time allotted. Hard task level trials require the subject to make 100 button presses, using their non-dominant pinky finger within 21 seconds to be successful. Easy task level trials require the subject to make 30 button presses, using their dominant index finger within 7 seconds. For easy task trials, subjects are eligible to win the same amount of money on each trail if they successfully complete the task. For hard task trials, subjects are eligible to win higher amounts, which vary per trial. Subjects are not guaranteed to win the reward if they complete the task, as only some hard task trials are 'win' trials, while others are 'lose' trials in which no money is won. To help subjects determine which trials are more likely to be 'win' trials, one of three accurate probability cues are presented at the beginning of each trial, for both easy and hard tasks: high probability of winning (88%), medium probability of winning (50%), and low probability of winning (12%). Equal proportions of each probability level across the experiment. Each level of probability appeared once in conjunction with each level of reward value for the hard task. Trials will be presented in the same randomized order to all subjects. All trials begin with a 1-second fixation cross, following a 5-second choice period in which subjects are presented with information regarding the probability of receiving a reward, and the reward magnitude of the hard task. Subjects are told that if they do not make a choice within 5 seconds, they will be randomly assigned to either an easy or hard task for that trial. After making a choice, subjects are then shown a 1-second Ready screen before the task begins. Following the task, subjects are shown a 2-second feedback screen stating whether the subject won money for that trial (reward feedback). In total, easy task trials take ~15 seconds to complete, while hard task trials take ~30 seconds. Subjects are told they will receive a base-rate compensation for their participation in the study overall. Additionally, all subjects are told that two of their 'win' trials would be randomly selected at the end of the experiment as 'incentive trials.' For these incentive trials, subjects will receive additional real monetary compensation. Subjects will be informed that they have twenty minutes to play as many trials as they can. Yet, since hard task trials take about twice as long to complete as the easy task trials, the number of trials each subject can play depends, in part, on the choices the subject makes. This means making the decision to complete more hard task trials in the beginning of the game could reduce the number of trials, and, in turn, may mean the subject does not get a chance to play the high-value/high-probability trials which might appear later in the game. This trade-off will be thoroughly explained to each subject, but subjects will not be given any information regarding the distribution of the trial types. The goal of this trade-off is to help ensure that neither strategizing by always choosing the easy trial, nor by always choosing the hard trial, could lead to an 'optimal' task performance. Moreover, the complexity of variables (varying monetary reward, probability, time pressure) does not lend itself to a formal calculation of an optimal response selection, and subjects are required to decide within a brief amount of time. This is done to help ensure that subject decisions reflect individual differences in willingness to expend effort for a given level of expected reward value.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria must be met for all subjects to be considered eligible to participate:

1. 18 years old or older
2. Equal numbers of men and women, as well as racial and ethnic makeup representative of surrounding area
3. Able to speak, read, and understand English
4. In generally stable health
5. Sign informed consent document

The following inclusion criteria must be met for chronic pain patients to be considered eligible to participate:

1. Patients must report chronic pain for more than 1 year.
2. The reported pain should be rated at ≥ 40/100

Exclusion Criteria:

General exclusion criteria for all subjects include:

1. Significant other medical disease, such as unstable diabetes mellitus, congestive heart failure, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy
2. History of traumatic brain injury (TBI)
3. Current misuse/dependence on substance(s), including alcohol, at the time of study enrollment
4. Major psychiatric disorder during the past 6 months
5. Significantly abnormal laboratory values, which include, but are not limited to, the following:

   1. White blood cell (WBC) < 1.5 or >15.0 x 10^3/μL
   2. Hemoglobin (Hgb) < 8 gm/dL
   3. Hematocrit (Hct) < 24% or > 50%
   4. Platelets (Plts) <50 or > 1000 x10^3
   5. Creatine > 2 mg/dL
   6. Glucose > 125 mg/dL
   7. Aspartate aminotransferase (AST) > 250 U/L
   8. Alanine Transaminase (ALT) > 250 U/L
   9. Bilirubin > 3 mg/dL
6. Intra-axial implants (e.g. - spinal cord stimulators or pumps)
7. Inability to adequately perform the finger-span visual tracking task (training for rotating pain perception, see Brain Imaging Details).
8. All MRI exclusionary criteria: any metallic implants, brain or skull abnormalities, tattoos on large body parts, pregnancy, and claustrophobia.
9. In the judgement of the investigator, unable or unwilling to follow the protocol and instructions.
10. Gambling addiction self-reported during screening process (ensure computer-based games do not cause psychological or emotional problems)
11. Chronic pain patients with past history of allergic reactions to methylphenidate or levodopa/carbidopa.

For healthy control subjects, current complaint(s) of pain, or a history of pain lasting >4 weeks in the last year, will be excluded from participating.

In addition, exclusion criteria for chronic pain subjects also includes:

1. Pain that is associated with any systemic signs or symptoms (e.g. - fever, chills)
2. Evidence of rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures, fibromyalgia, history of tumor(s) in the back.
3. Involvement in litigation regarding their pain, or having a disability claim, or receiving workman's compensation, or seeking either because of their pain.
4. Treated with methadone for opioid use disorder (i.e. - not just for pain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
mean change in amygdala volume | baseline to 3 hours
  Amygdala volume will be measured using T1w MPRAGE structural images. The mean change in amygdala volume will be the volume of amygdala before administering the drug or placebo minus the volume of amygdala after administering the drug or placebo.
mean change in hippocampus volume | baseline to 3 hours
  Hippocampus volume will be measured using T1w MPRAGE structural images. The mean change in hippocampus volume will be the volume of hippocampus before administering the drug or placebo minus the volume of hippocampus after administering the drug or placebo.
mean change in thalamus volume | baseline to 3 hours
  Thalamus volume will be measured using T1w MPRAGE structural images. The mean change in thalamus volume will be the volume of thalamus before administering the drug or placebo minus the volume of thalamus after administering the drug or placebo.
mean change in Nucleus accumbens volume | baseline to 3 hours
  Nucleus accumbens volume will be measured using T1w MPRAGE structural images. The mean change in Nucleus accumbens volume will be the volume of Nucleus accumbens before administering the drug or placebo minus the volume of Nucleus accumbens after administering the drug or placebo.
mean change in amygdala activity | baseline to 3 hours
  Amygdala activity will be determined using Blood Oxygen Level Dependent (BOLD) fMRI sequences. The mean change in amygdala activity will be the activity of amygdala before administering the drug or placebo minus the activity of amygdala after administering the drug or placebo.
mean change in hippocampus activity | baseline to 3 hours
  Hippocampus activity will be determined using Blood Oxygen Level Dependent (BOLD) fMRI sequences. The mean change in hippocampus activity will be the activity of hippocampus before administering the drug or placebo minus the activity of hippocampus after administering the drug or placebo.
mean change in thalamus activity | baseline to 3 hours
  Thalamus activity will be determined using Blood Oxygen Level Dependent (BOLD) fMRI sequences. The mean change in thalamus activity will be the activity of thalamus before administering the drug or placebo minus the activity of thalamus after administering the drug or placebo.
mean change in Nucleus Accumbens activity | baseline to 3 hours
  Nucleus Accumbens activity will be determined using Blood Oxygen Level Dependent (BOLD) fMRI sequences. The mean change in Nucleus Accumbens activity will be the activity of Nucleus Accumbens before administering the drug or placebo minus the activity of Nucleus Accumbens after administering the drug or placebo.

SECONDARY OUTCOMES:
Effort Expenditure for Reward Task (EEfRT) | baseline to 3 hours
  This is a multi-trial task where subjects are given an opportunity on each trial to choose between two different task difficulty levels associated with varying levels of monetary reward. Each trial presents the subject with a choice between, a 'hard task' ((high cost/high reward (HC/HR) and an 'easy task' (low cost/low reward (LC/LR)) option, which require different amounts of speeded manual button pressing. For easy-task choices, subjects are eligible to win the same amount on each trial if they successfully complete the task. For hard-task choices, subjects are eligible to win higher amounts that vary per trial. Performance on EEfRT is modulated by mesolimbic dopamine transmission which is well known to be altered in chronic pain, and in MDD39. The responses are scored from 0 - 1 as proportions of high cost/high rewards tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No